CLINICAL TRIAL: NCT02029235
Title: Post-operative Analgesia in Elective, Soft-tissue Hand Surgery: A Randomized, Double Blind Comparison of Acetaminophen/Ibuprofen Versus Acetaminophen/Hydrocodone
Brief Title: Post-operative Analgesia in Elective, Soft-tissue Hand Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination due to slower than anticipated recruitment.
Sponsor: Alexander Payatakes, M.D. (Other)
Responsible Party: Sponsor-Investigator, Alexander Payatakes, M.D., Principal Investigator / Sponsor, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB - 00076
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Carpal Tunnel; Ganglion Cyst; Trigger Finger; De Quervain Disease
Keywords: Adult; soft-tissue hand surgery
MeSH Terms: conditions — Median Neuropathy; Ganglion Cysts; Trigger Finger Disorder; De Quervain Disease | interventions — Acetaminophen; Ibuprofen; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen/Ibuprofen (AIBU) Group (Active Comparator): Acetaminophen 500 mg and Ibuprofen 400 mg
  Interventions: Drug: Acetaminophen/Ibuprofen
- Acetaminophen/Hydrocodone (AH) Group (Active Comparator): Acetaminophen 325 mg and Hydrocodone 5 mg
  Interventions: Drug: Acetaminophen/Hydrocodone

INTERVENTIONS:
Drug: Acetaminophen/Ibuprofen — Postoperatively, subjects will be given acetaminophen 500 mg / ibuprofen 400mg every 4 hours, as needed, for one week or until essentially pain-free
  Other Names: Acetaminophen/Tylenol; Ibuprofen/Advil/Motrin
  Arms: Acetaminophen/Ibuprofen (AIBU) Group
Drug: Acetaminophen/Hydrocodone — Postoperatively, subjects will be given acetaminophen 325 mg / hydrocodone 5 mg every 4 hours, as needed, for one week or until essentially pain-free
  Other Names: Norco
  Arms: Acetaminophen/Hydrocodone (AH) Group

SUMMARY:
The purpose of this research study is to find out which combination of pain medications following surgery work the best and result in the fewest side effects.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind study comparing the efficacy of acetaminophen/hydrocodone (AH) to acetaminophen/ibuprofen (AIBU) in providing adequate post-operative pain relief in elective, soft tissue hand surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Male or Female (non-pregnant)
* Elective, soft tissue hand surgery indicated based on diagnosis made by either clinical exam or diagnostic studies (ie nerve conduction study, EMG) or a combination of the two (carpal tunnel release, trigger finger release, first dorsal compartment release, ganglion cyst excision, second extensor compartment release)
* Subjects are capable of giving informed consent

Exclusion Criteria:

* Allergy to study medication
* Any pre-existing pain condition requiring analgesia
* Fibromyalgia
* Recent upper gastrointestinal bleeding
* Coagulopathy (primary or medication-related)
* Renal impairment
* Liver disease
* Pregnancy
* Patients who consent to the study but require unexpected admission, including those requiring admission resulting from operative complications, will be excluded before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Payatakes, M.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodgers J, Cunningham K, Fitzgerald K, Finnerty E. Opioid consumption following outpatient upper extremity surgery. J Hand Surg Am. 2012 Apr;37(4):645-50. doi: 10.1016/j.jhsa.2012.01.035. Epub 2012 Mar 10. PMID 22410178
- [Background] Kuehn BM. Opioid prescriptions soar: increase in legitimate use as well as abuse. JAMA. 2007 Jan 17;297(3):249-51. doi: 10.1001/jama.297.3.249. No abstract available. PMID 17227967
- [Background] Centers for Disease Control and Prevention (CDC). Emergency department visits involving nonmedical use of selected prescription drugs - United States, 2004-2008. MMWR Morb Mortal Wkly Rep. 2010 Jun 18;59(23):705-9. PMID 20559200
- [Background] Mitchell A, McCrea P, Inglis K, Porter G. A randomized, controlled trial comparing acetaminophen plus ibuprofen versus acetaminophen plus codeine plus caffeine (Tylenol 3) after outpatient breast surgery. Ann Surg Oncol. 2012 Nov;19(12):3792-800. doi: 10.1245/s10434-012-2447-7. Epub 2012 Jun 20. PMID 22713999
- [Background] White PF, Tang J, Wender RH, Zhao M, Time M, Zaentz A, Yumul R, Sloninsky A, Naruse R, Kariger R, Webb T, Fermelia DE, Tsushima GK. The effects of oral ibuprofen and celecoxib in preventing pain, improving recovery outcomes and patient satisfaction after ambulatory surgery. Anesth Analg. 2011 Feb;112(2):323-9. doi: 10.1213/ANE.0b013e3182025a8a. Epub 2010 Dec 14. PMID 21156974
- [Background] Beauregard L, Pomp A, Choiniere M. Severity and impact of pain after day-surgery. Can J Anaesth. 1998 Apr;45(4):304-11. doi: 10.1007/BF03012019. PMID 9597202
- [Background] Dexter F, Chestnut DH. Analysis of statistical tests to compare visual analog scale measurements among groups. Anesthesiology. 1995 Apr;82(4):896-902. doi: 10.1097/00000542-199504000-00012. PMID 7717561

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited during clinic visits to discuss elective, soft tissue hand surgery at a single academic medical center between February 2015 and October 2017. The first participant was enrolled in February 2015, and the last participant was enrolled in October 2017.
Pre-assignment Details: Seven patients withdrew or were excluded prior to randomization due to cancellation of surgery (3), refusal to participate (3), and a newly diagnosed gastrointestinal ulcer (exclusion criterion) prior to surgery (1).
Groups:
- Acetaminophen/Ibuprofen (AIBU) Group: Postoperatively, subjects were given:
  Acetaminophen 500 mg / Ibuprofen 400 mg every 4 hours, as needed, for one week or until essentially pain-free.
- Acetaminophen/Hydrocodone (AH) Group: Postoperatively, subjects were given:
  Acetaminophen 325 mg / Hydrocodone 5 mg every 4 hours, as needed, for one week or until essentially pain-free.
Period: Overall Study
Arm/Group | Acetaminophen/Ibuprofen (AIBU) Group | Acetaminophen/Hydrocodone (AH) Group
Started | 34 | 31
Completed | 30 | 30
Not Completed | 4 | 1
Not completed — Non-compliance with study meds or diary | 4 | 1

BASELINE CHARACTERISTICS:
Population: Subjects randomized into study groups and completing protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen/Ibuprofen (AIBU) Group | Acetaminophen/Hydrocodone (AH) Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Full Range); unit: years] | 52 [18 to 86] | 53 [18 to 75] | 53 [18 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 12 | 13 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Patient Health Questionnaire (PHQ-9) [Mean (Full Range); unit: units on a scale (total score)] — The Patient Health Questionnaire (PHQ-0) objectifies degree of depression severity.
  It provides a total score on a scale of 0 - 27, with higher being worse (i.e. more severe depression).
  units on a scale (total score) | 1.83 [0 to 12] | 2.63 [0 to 14] | 2.23 [0 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Comparison of Pain Intensity Level
Description: Subjects asked to fill out a patient diary recording their pain intensity level (on 100mm Visual Analog Scale) prior to taking study medication every 4 hours.
  The daily average pain intensity levels are reported as a score on a scale of 0-100, with higher score meaning worse outcome.
  The daily average pain levels were assessed daily for 1 week post-operatively, then compared between the 2 groups using a two-group Student's t-test.
Time Frame: 1 week post-operatively
Measure: Mean (Full Range); unit: score on a scale (0-100, higher = worse)
Arm/Group | Acetaminophen/Ibuprofen (AIBU) Group | Acetaminophen/Hydrocodone (AH) Group
Number analyzed (Participants) | 30 | 30
score on a scale (0-100, higher = worse)
  Daily average pain intensity level on PostOp Day 1 | 22.17 [0 to 100] | 24.07 [0 to 100]
  Daily average pain intensity level on PostOp Day 2 | 22.22 [0 to 93] | 30.16 [0 to 95]
  Daily average pain intensity level on PostOp Day 3 | 15.67 [0 to 75] | 22.11 [0 to 90]
  Daily average pain intensity levelon PostOp Day 4 | 13.17 [0 to 55] | 18.53 [0 to 90]
  Daily average pain intensity level on PostOp Day 5 | 14.03 [0 to 67] | 16.61 [0 to 90]
  Daily average pain intensity level on PostOp Day 6 | 13.44 [0 to 50] | 13.58 [0 to 73]
  Daily average pain intensity level on PostOp Day 7 | 12.67 [0 to 65] | 13.00 [0 to 63]
Statistical Analysis 1: Comparison: Acetaminophen/Ibuprofen (AIBU) Group vs Acetaminophen/Hydrocodone (AH) Group; Null hypothesis: No difference between groups Power analysis: A sample size of 16 in each group had an 80% power to detect a difference in means of 10 mm; Test type: Other; p = 0.24, t-test, 2 sided

2. Secondary Outcome: Efficacy Comparison of Pain Relief
Description: Subjects asked to fill out a patient diary recording their pain relief (on a Likert scale) one hour after taking study medication every 4 hours.
  Daily average pain relief scores are reported as a score on a scale of 0-3, with higher score meaning better outcome.
  The daily average pain relief scores were assessed daily for 1 week post-operatively, then compared using generalized linear mixed-effects models
Time Frame: 1 week postoperatively
Measure: Mean (Full Range); unit: score on a scale (0-3, higher = better)
Arm/Group | Acetaminophen/Ibuprofen (AIBU) Group | Acetaminophen/Hydrocodone (AH) Group
Number analyzed (Participants) | 30 | 30
score on a scale (0-3, higher = better)
  Daily average pain relief on PostOp Day 1 | 1.84 [1 to 3] | 1.53 [1 to 3]
  Daily average pain relief on PostOp Day 2 | 2.27 [1 to 3] | 1.76 [1 to 3]
  Daily average pain relief on PostOp Day 3 | 2.63 [1 to 3] | 2.33 [1 to 3]
  Daily average pain relief on PostOp Day 4 | 2.91 [1 to 3] | 2.46 [1 to 3]
  Daily average pain relief on PostOp Day 5 | 2.88 [1 to 3] | 2.54 [1 to 3]
  Daily average pain relief on PostOp Day 6 | 2.87 [1 to 3] | 2.84 [1 to 3]
  Daily average pain relief on PostOp Day 7 | 2.96 [1 to 3] | 2.88 [1 to 3]
Statistical Analysis 1: Comparison: Acetaminophen/Ibuprofen (AIBU) Group vs Acetaminophen/Hydrocodone (AH) Group; Null hypothesis: No difference between groups; Test type: Other; p = 0.06, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Definition consistent with those listed on clinicaltrials.gov website.
  Adverse event collection occurred at postop day 7 phone call, as well as first follow-up clinic-visit.
Arm/Group | Acetaminophen/Ibuprofen (AIBU) Group | Acetaminophen/Hydrocodone (AH) Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 1/34 | 7/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen/Ibuprofen (AIBU) Group (N=34) | Acetaminophen/Hydrocodone (AH) Group (N=31)
Drowsiness (Nervous system disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to slower than anticipated recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT02029235/Prot_SAP_000.pdf